CLINICAL TRIAL: NCT04909424
Title: Prevalence of Cutaneous Enterococci at Femoral Insertion Site in Transcatheter Aortic Valve Implantation (TAVI)
Acronym: Entero-TAVI
Status: Completed | Type: Observational
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Dr Benoit Fontenel, Principal investigator, MD, Clinique Pasteur
Other Study IDs: 2021-A00370-41
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease
Keywords: Enterococci; Infective endocarditis; Antibiotic prophylaxis; TAVI
MeSH Terms: conditions — Aortic Valve Disease; Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general rules of antibiotic prophylaxis in surgery or interventional medicine include the choice of an antibiotic active on the bacteria most frequently encountered in surgical site infections. This antibiotic must cover, the bacteria present on the skin and recognized as responsible for surgical site infections.

The aim of this study is to identify bacteria found in skin flora in the inguinal region of patients undergoing Transcatheter Aortic Valve Implantation (TAVI). Flora found will allow to evaluate the impact of skin preparation and antibiotic prophylaxis protocols as they are currently practiced.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for aortic valve replacement by TAVI procedure with trans femoral approach
* Patient with pre-TAVI assessment performed at Clinique Pasteur
* Patient affiliated or beneficiary of a social security scheme
* Patient accepting to participate and having given his no objection

Exclusion Criteria:

* TAVI procedure by non-trans femoral approach
* Protected patients: Adults under guardianship or other legal protection; Pregnant or breastfeeding woman; Hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In hospital patients for pre TAVI assessment at Clinique Pasteur
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Enterococci prevalence | At Day 0 at TAVI intervention time (preoperative)
  Proportion of patients with Enterococcus feacalis and other Enterococci in inguinal flora before TAVI

SECONDARY OUTCOMES:
Skin flora of the groin | At Day 0 at TAVI intervention time (preoperative) before skin disinfection
  Bacteria profile of inguinal skin
Skin flora of the groin | At Day 0 at TAVI intervention time (preoperative) after skin disinfection
  Bacteria profile of inguinal skin
Infectious events | From day of TAVI to 1 year after intervention
  Occurrence of infective endocarditis or other infectious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bonnet, MD, Study Chair — Clinique Pasteur; Nicolas Combes, MD, Study Chair — Clinique Pasteur; Benoit Fontenel, MD, Study Chair — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France